## Document related to the research project:

## Long-term Survivors of High-grade glioma

Review Committee of the Capital Region of Denmark (H-16035446) and the Danish Data Protection Agency (2012-58-0004).







Karin Piil, BSC, Master of Health Science, Nursing, Ph.D. The University Hospitals Center for Health Research (UCSF) and the Center for Integrated Rehabilitation of Cancer Patients (CIRE) in collaboration with the Neuro-Oncology team, Rigshospitalet. Email: <a href="mailto:Karin.piil@regionh.dk">Karin.piil@regionh.dk</a>

Mary Jarden, Senior Researcher, Associate Professor, cand. cur., Ph.D. University Hospitals Center for Health Research (UCSF), Rigshospitalet, Center for Integrated Rehabilitation of Cancer Patients (CIRE) and University of Copenhagen.

Statistical analysis The PS, the The Hospital Anxiety and Depression Scale (HADS) sub-scales, the The Functional Assessment of Cancer Therapy, General and brain cancer (FACT-G and FACT-Br) sub-scales and the responses to the ordinal items of the leisure time physical activity scale will be analysed separately. Socio-economic information and data from questionnaires will be entered into a database. The questionnaires will be analyzed according to their manuals.

Categorical variables will be reported as frequencies and percentages, while continuous variables are reported as mean and standard deviations (s.d.) using a significance level of p\0.05. HADS and FACT-Br data refer to the normative values. The statistical analysis will be performed with SAS (Statistical Analysis System) statistical software, version 9.3.